CLINICAL TRIAL: NCT06744712
Title: Pharmacogenomic Testing in Pediatric Hematology/Oncology Patients
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Wake Forest University Health Sciences (Other)
Collaborators: Atrium Health Levine Cancer Institute (Other); OneOme, LLC (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Supportive Care
Other Study IDs: IRB00104368; LCI-PED-NDPO-PGx-001 (Other: Atrium Health); NCI-2025-00567 (Other: National Cancer Institute)
Record Dates: First submitted 2024-11-27; First posted 2024-12-20 (Actual); Last update posted 2026-01-07 (Actual); Status verified 2026-01

CONDITIONS: Pediatric Cancer
Keywords: Pharmacogenomic; Anti-Cancer Therapy
MeSH Terms: conditions — Neoplasms | interventions — Pharmacogenomic Testing

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Pharmacogenomic (PGx) Testing (Experimental)
  Interventions: Other: Pharmacogenomic Testing

INTERVENTIONS:
Other: Pharmacogenomic Testing — Pharmacogenomic testing will be completed by the vendor. The vendor is certified under CLIA-88 and accredited by the College of American Pathologists as qualified to perform high-complexity testing. Genomic DNA extracted from the swab will be analyzed by PCR using Thermo Fisher TaqMan® and/or LGC Biosearch BHQ® probe-based methods to interrogate the variant locations listed in (See Appendix II). Twenty-seven genes are evaluated and reported.

SUMMARY:
Pharmacogenomic (PGx) testing involves analyzing variants of genes associated with drug metabolism, transport and medication targets. PGx testing uses an individual's genetic factors, such as single nucleotide polymorphisms (SNPs), to personalize therapy or dose a selection of medications. PGx testing has traditionally been used to test single genes, but there are now platforms allowing a panel of genes to be tested at once. To date there has not been a comprehensive screening of pediatric oncology patients to determine the prevalence of genetic variants that may affect anticancer therapy and supportive care medications. This study would allow us to summarize the frequency of clinically relevant gene-drug interactions and actionable genetic polymorphisms in pediatric oncology patients.

DETAILED DESCRIPTION:
This is a prospective, non-treatment, interventional single-arm study evaluating PGx results and modifications made to anticancer therapy and supportive medication administration based on PGx results in participants ≤ 26 years old with a newly diagnosed malignancy or bone marrow transplant candidate with non-malignant diagnosis who has not yet undergone myeloablative conditioning regimen.

Potential candidates will be presented with consent. Patients who agree will undergo the informed consent process, and participants who consent will be screened for eligibility. Those meeting eligibility criteria will be enrolled and undergo buccal swab collection. The buccal swab will be collected and sent for PGx testing at time of enrollment.

A copy of the test results in PDF (Portable Document Format) format and PGx consultation note will be uploaded to the participant's electronic medical record (EMR) and will be available to the participant via the MyAtrium Patient Portal and treating oncologist in the EMR. Results will also be reviewed by the pediatric oncology pharmacists. Apart from the availability and use of PGx test results to guide pharmacotherapy, participants will receive standard of care treatment as recommended by their primary oncologist.

During study participation, dose modifications made to anticancer therapy and supportive care medications based on PGx results will be collected every three months.

Participants are enrolled voluntarily after informed consent/assent and will not be reimbursed for study participation. Participants will receive PGx testing at no cost.

ELIGIBILITY:
Inclusion Criteria:

1. Written informed consent and HIPAA authorization for release of personal health information, and assent when applicable, from the participant, parent or legal guardian.
2. Age ≤ 26 years at the time of consent.
3. Newly diagnosed with a malignancy and planning to undergo anti-cancer therapy; or bone marrow transplant candidate with a non-malignant diagnosis who has not yet undergone myeloablative conditioning regimen.

Exclusion Criteria:

1. Anti-cancer therapy has already been initiated. Note: Enrollment after initiation of intrathecal chemotherapy will be allowed.
2. Previously received bone marrow transplant or planning to receive as part of initial upfront therapy for a malignant condition.
3. Prior history of tissue or organ transplant.

Max Age: 26 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 130 (Estimated)
Dates: Start 2026-03 (Estimated); Primary Completion 2027-08 (Estimated); Study Completion 2028-07 (Estimated)

PRIMARY OUTCOMES:
Gene-drug interaction | 3, 6, 9, 12 months after enrollment
  A gene-drug interaction occurs when an individual carrying a variant form of a gene is administered a drug that serves as a substrate for the enzyme or transporter encoded by that gene. Clinically relevant gene-drug interactions are defined in the CPIC (Clinical Pharmacogenetics Implementation Consortium) guidelines or the FDA Table of Pharmacogenomic Associations. Gene-drug interaction is a binary variable (interaction present or interaction absent). Each clinically relevant gene-drug interaction from the pharmacogenomic testing will be reported.
Genotype | Baseline
  Genes involved in toxicity and efficacy of pediatric anticancer therapy and supportive care medications, as listed in CPIC or FDA Table of Pharmacogenomic Association guidelines, are tested for genetic polymorphisms using the OneOme RightMed Comprehensive Test. Each gene's genotype is classified as a binary variable (actionable or not actionable).

SECONDARY OUTCOMES:
Anticancer treatment modification based on PGx test result | 3, 6, 9, 12 months after enrollment
  Anticancer treatment modification includes modifications in medication, dosage, or treatment frequency. Anti-cancer therapy treatment modification is a binary variable (yes or no), where 'yes' indicates that at least one type of modification occurred.
Modification in supportive medication based on PGx test result | 3, 6, 9, 12 months after enrollment
  Modification in supportive medication includes modifications in medication, dosage, treatment frequency, or adding new medication. Modification in supportive medication is a binary variable (yes or no), with 'yes' indicates at least one type of modification occurred.

CONTACTS AND LOCATIONS:
Overall Officials: Erin Trovillion, MD, Principal Investigator — Wake Forest University Health Sciences
Locations (1):
- Levine Childrens Hospital Pediatric Cancer and Blood Disorders, Charlotte, North Carolina, United States